CLINICAL TRIAL: NCT06684535
Title: Role of Dexmedetomidine as an Adjuvant in External Oblique Intercostal Plane Block for Post Thoracotomy Pain: A Randomized Controlled Trial
Brief Title: Dexmedetomidine as an Adjuvant in External Oblique Intercostal Plane Block for Post Thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR904/10/24
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Dexmedetomidine; Adjuvant; External Oblique Intercostal Plane Block; Thoracotomy; Pain
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients will receive 29 ml bupivacaine 0.25% + 1 ml dexmedetomidine 0.5 μg/kg.
  Interventions: Drug: Dexmedetomidine
- Control group (Active Comparator): Patients will receive 29 ml bupivacaine 0.25% + 1 ml saline.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive 29 ml bupivacaine 0.25% + 1 ml dexmedetomidine 0.5 μg/kg.
  Arms: Dexmedetomidine group
Drug: Saline — Patients will receive 29 ml bupivacaine 0.25% + 1 ml saline.
  Arms: Control group

SUMMARY:
This study aims to evaluate the role of dexmedetomidine as an adjuvant in external oblique intercostal plane block for post-thoracotomy pain.

DETAILED DESCRIPTION:
External oblique intercostal plane block (EOIPB) is a novel block that has been described as an important modification of the fascial plane blocks that can consistently involve the upper lateral abdominal walls.

Dexmedetomidine is a selective alpha 2- adrenoceptor agonist possessing sedative, anxiolytic, and analgesic properties without the development of respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Scheduled for open thoracotomy.

Exclusion Criteria:

* Patients with neurological or intellectual disability.
* Infection at the injection site.
* Drug abuse.
* Allergic reaction to local anesthetics.
* Coagulation abnormalities.
* Pregnancy.
* Body Mass Index (BMI) ≥35 kg/m2.
* Severe cardiovascular problems.
* Diabetic neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated) will be recorded.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline.
Total morphine consumption | 48 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4.
Degree of pain | 48 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.
Heart rate | Every 15 min till the end of surgery
  Heart rate will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Mean arterial pressure | Every 15 min till the end of surgery
  Mean arterial pressure will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Incidence of adverse events | 48 hours postoperatively
  Incidence of adverse events such as pneumothorax, local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.